CLINICAL TRIAL: NCT07022067
Title: EVOLVING AZIMUTH IN MUSA CONTEXT
Acronym: AZIMUSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: ASST Grande Ospedale Metropolitano Niguarda (Other); University of Milan (Other)
Responsible Party: Principal Investigator, Stefano Carugo, Director of the Department of Cardio-Thoracic-Vascular Diseases, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4372
Record Dates: First submitted 2025-05-14; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure; Blood Pressure; Weight Change; Telemonitoring
MeSH Terms: conditions — Heart Failure; Body Weight Changes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): The patient in the experimental arm downloads a telemonitoring application where they enter their pressure and body weight data, which is revised by the hospital team via a platform. The patient complete a questionnaire during enrollment and during two follow-ups (3 months and 6 months) to examine various dimensions.
  Interventions: Device: Telemonitoring app
- Standard care (No Intervention): The patient in the standard care arm do not downloads a telemonitoring application, but they continue with normal medical indication. The patient complete a questionnaire during enrollment and during two follow-ups (3 months and 6 months) to examine various dimensions.

INTERVENTIONS:
Device: Telemonitoring app — periodic measurement of blood pressure and body weight
  Arms: Telemonitoring

SUMMARY:
Non-pharmacological, randomized, nonprofit medical device intervention. The study aims to identify the positive impacts (co-creation), and negative impacts (co-destruction), resulting from the use of telemedicine, and, in particular, the telemonitoring service for patients with heart failure

DETAILED DESCRIPTION:
The patient diagnosed with heart failure is randomized to either the experimental or control arm. The patient in the experimental arm downloads a telemonitoring application where they enter their pressure and body weight data, which is revised by the hospital team via a platform. Patients from both arms complete a questionnaire during enrollment and during two follow-ups (3 months and 6 months) to examine various dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with chronic CS according to the ESC guidelines;
* Over 18 years of age;
* Patients admitted to hospital or with access to first aid within the last year;
* Smartphome that meets the digital requirements (ie Android or iOS able to download and use the application);
* Wi-Fi or 3G coverage at home;
* Ability to give written informed consent.

Exclusion Criteria:

* Severe psychiatric disorder
* Inability to use portable technologies
* Patients unable to use the equipment provided
* Patients who deny consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
PAM13-I | 6 months
  The Patient Activation Measure (PAM13-I) is a brief, validated instrument that assesses patient knowledge, skills, and confidence for disease self-management. It consists of 13 items on a Likert scale. According to the American version of PAM 13, each item has five response categories with scores from 1 to 5: (1) "Strongly Disagree", (2) "Disagree", (3) "Agree", (4) "Strongly Agree" and (5) "Not Applicable". The instrument design reflects the four stages of activation in a progressing difficulty of the items: level 1 (patients believe that their role is important: items 1 and 2), level 2 (patients have confidence and knowledge to take action: items 3-8) level 3 (taking action: items 9-11) and level 4 (staying on course under stress: items 12 and 13).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Prof. Carugo, Principal Investigator — IRCCS Fondazione Caì Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy, Italy